CLINICAL TRIAL: NCT03699085
Title: A Longitudinal Collaborative Care Model for Patients With Opioid Problems: Emergency Department Longitudinal Integrated Care (ED-LINC)
Brief Title: Emergency Department Longitudinal Integrated Care
Acronym: ED-LINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lauren Whiteside, Assistant Professor, School of Medicine: Department of Emergency Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005447; K23DA039974 (NIH)
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Opioid-use Disorder; Emergency Department
Keywords: Opioid Use; Emergency Department; Collaborative Care
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals on the study team designated to conduct follow up interviews will be blinded to which arm participants belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED-LINC Intervention Condition (Experimental): Patients in this arm will receive the ED-LINC intervention. Elements of ED-LINC are based on evidence-based treatments and are central components of collaborative care. ED-LINC will be supported by a novel Emergency Department Information Exchange (EDIE) technology platform that allows for the creation of ED care plans and electronic alerts and will assist in care coordination of this complex population.
  Interventions: Behavioral: ED-LINC
- Usual Care Condition (No Intervention): Patients in this arm may receive a spectrum of consulting services visits including social work services, psychiatric consultation, inpatient psychiatry consult, rehabilitation psychology consultation, addiction intervention services, pain team consultation services that include MD psychiatric and PhD psychologist providers, spiritual care or other consulting services which shall count as usual care.

INTERVENTIONS:
Behavioral: ED-LINC — ED-LINC will include 1) A brief negotiated interview at the bedside with an emphasis on motivation to link to services 2) Pharmacotherapy including a discussion of opioid safety, take-home naloxone and initiation of buprenorphine from the ED for participants that are interested and eligible; 3) Longitudinal care management which will proceed for 3-months; and 4) Care plan in the Emergency Department Information Exchange (EDIE) system. This will be coupled with a study cell phone and a weekly supervisory case conference which is consistent with collaborative care principles.
  Arms: ED-LINC Intervention Condition

SUMMARY:
The overarching goal of this investigation is to develop and determine the feasibility of a multi-component intervention adapted from a collaborative care framework initiated in the ED for patients at risk for opioid use disorder. This study will provide important feasibility information for future studies of ED-LINC. The collaborative care intervention (ED-LINC) will be supported by a novel Emergency Departement (ED) health information exchange platform.

DETAILED DESCRIPTION:
The overarching goal of this investigation is to develop and determine the feasibility of a multi-component intervention adapted from a collaborative care framework initiated in the ED for patients at risk for opioid use disorder. According to the 2015 national survey on drug use and health, an estimated 3.8 million individuals over 12 years of age were currently misusing opioid pain relievers. An additional 329,000 people use heroin. The Emergency Department (ED) is currently at the forefront of this public health emergency and often a place where patients come for treatment of overdose and for treatment of medical problems related to illicit opioid use.

Overall, the goal is to establish the feasibility of a multi-component intervention called 'Emergency Department Longitudinal Integrated Care (ED-LINC)' which is guided by principles of collaborative care and is comprised of components that are evidence-based. ED-LINC is initiated from the ED and continues longitudinally for patients at-risk for opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Patients with at least one risk factor for opioid use disorder via the EMR pre-screen
* Patients with score of ≥ 4 on the NIDA modified ASSIST for illicit opioids (e.g. heroin) OR a score of ≥ 4 on the NIDA modified ASSIST for prescription opioids
* Currently have a phone
* Able to provide a phone number and one additional piece of contact information

Exclusion Criteria:

* They are incarcerated or under arrest
* Non-English speaking
* Live beyond a 50 mile radius of HMC
* Require active resuscitation in the ED or other clinical area at the time of RA approach
* Are receiving palliative care services or hospice care for a chronic illness such as metastatic cancer
* Are in the ED or hospital for a primary psychiatric emergency such as suicidal ideation or attempt
* Receiving chronic opioid therapy (COT) defined as prescription opioids for most days out of the last 90 days for a chronic pain condition
* In the ED for sexual assault

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Whiteside, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whiteside LK, Huynh L, Morse S, Hall J, Meurer W, Banta-Green CJ, Scheuer H, Cunningham R, McGovern M, Zatzick DF. The Emergency Department Longitudinal Integrated Care (ED-LINC) intervention targeting opioid use disorder: A pilot randomized clinical trial. J Subst Abuse Treat. 2022 May;136:108666. doi: 10.1016/j.jsat.2021.108666. Epub 2021 Nov 24. PMID 34952745

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Baseline survey completed prior to randomization
Period: Overall Study
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.7) | 39.4 (9.3) | 37.4 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 11 | 12 | 23
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Heroin Use [Count of Participants; unit: Participants] — Self reported heroin use in past 30 days of assessment
  Participants | 19 | 19 | 38
Prescription Opioid Misuse [Count of Participants; unit: Participants] — Self reported prescription opioid misuse in prior 30 days before assessment
  Participants | 6 | 2 | 8
Lifetime Opioid Overdose [Count of Participants; unit: Participants] — Percentage of participants with self reported history of opioid overdose in lifetime
  Participants | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Refusal Rate
Description: Percentage of subjects who agree to participate in screening survey prior to determining eligibility status. Potential subjects identified by suspected risky substance use history based on EMR review
Time Frame: Baseline
Population: Potential subjects identified by suspected history of risky substance use based on EMR review
Measure: Count of Participants; unit: Participants
Groups:
- Approached Subjects: Number of potential subjects who were approached for potential participation
Arm/Group | Approached Subjects
Number analyzed (Participants) | 118
Participants
  Refused Screening Survey | 5
  Participated in Screening Survey | 113

2. Primary Outcome: Follow up Completion Rates
Description: The number of participants who completed follow-ups at 6 month time point.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
Number analyzed (Participants) | 20 | 20
Participants
  Completed 6 month followup | 18 | 19
  No 6 month followup | 2 | 1

3. Primary Outcome: ED-LINC Intervention and Usual Care Process Outcomes
Description: Number of participants that received at least 1 ED-LINC element
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
Number analyzed (Participants) | 20 | 20
Participants
  At least 1 ED LINC element received | 20 | 0
  No ED LINC elements received | 0 | 20

4. Primary Outcome: Implementation Appropriateness
Description: Participants randomized to ED-LINC care were asked about the appropriateness of interventional activities.by rating the agreeability of the statement "ED LINC seemed fitting and suitable"
Time Frame: 6 months
Population: Participants were asked to rate the agreeability of the statement "ED LINC seemed fitting and suitable"
Measure: Count of Participants; unit: Participants
Arm/Group | ED-LINC Intervention Condition
Number analyzed (Participants) | 20
Participants
  Agreed or Completely Agreed | 18
  Answered OTHER than Agreed or Completely Agreed | 2

5. Primary Outcome: ED-LINC Satisfaction
Description: Client Satisfaction Questionnaire (CSQ-8) questions (8-32) will be used to assess satisfaction with ED-LINC, in which greater numbers designate higher satisfaction (32 is maximum or highest satisfaction rating possible)
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
Number analyzed (Participants) | 20 | 20
score on a scale | 29 [26 to 32] | 30 [26 to 32]

6. Primary Outcome: Perception of Care Coordination
Description: The Patient Assessment of Chronic Illness Care - Coordination (PACIC-C) questions will be asked of all participants, where greater numbers indicate perception was more coordinated (greater number is better). For the scale, scores must be discrete numbers, with a minimum possible value of 5 and maximum possible value of 25.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
Number analyzed (Participants) | 18 | 19
score on a scale | 15 [11.25 to 19.25] | 13 [9 to 15.5]
Statistical Analysis 1: Comparison: ED-LINC Intervention Condition vs Usual Care Condition; Wilcoxon rank-sum test is used, which ranks the values in each group, sums the ranks and determines the probability that they are the same. The probability p-value is reported; Test type: Equivalence — A p value of < 0.05 suggests the groups are different; p = 0.38, Wilcoxon (Mann-Whitney) — A p value of < 0.05 suggests the groups are different

7. Secondary Outcome: Substance Use
Description: Comparison between control population and intervention population based on substance use measured utilizing a time-line follow back (TLFB) calendar administered by the research assistant to for past 30-day heroin use at TLFB timepoints (Baseline, 1 month, 3 months, 6 months). Table shows the average of unadjusted TLFB days of Heroin Use with 95% Confidence Interval.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: unadjusted TLFB days
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
Number analyzed (Participants) | 20 | 20
unadjusted TLFB days
  Baseline | 18.3 (2.89) | 16.85 (2.80)
  Month 1 | 11.95 (2.95) | 12.85 (2.93)
  Month 3 | 8.9 (2.88) | 12.45 (3.13)
  Month 6 | 13.1 (2.92) | 9.4 (3.06)
Statistical Analysis 1: Comparison: ED-LINC Intervention Condition vs Usual Care Condition; Comparison of control and intervention populations based on substance use measured utilizing a time-line follow back (TLFB) calendar administered by the research assistant to for past 30-day heroin use. This is a covariate-adjusted mixed effects regression model at TLFB timepoint of 6 months. A number greater than 1.0 indicates a higher incidence of heroin use in the past 30 days at the 6 month timepoint for intervention group compared to control group; Test type: Superiority — Adjusted mixed effects regression models were used to determine whether patients in the intervention and control group manifested different patterns of change in days of heroin use in the past 30 days in terms of incidence-rate ratio. We applied a negative binomial distribution to help account for overdispersion of outcome data; p = 0.68, Regression, Cox — A p value of < 0.05 suggests the groups are different; Incidence rate ratio = 1.29, 95% CI 2-sided [0.38 to 4.37] — A number greater than 1.0 indicates a higher incidence rate of heroin use in past 30 days for intervention group compared to control group

8. Secondary Outcome: Health Care Utilization
Description: Emergency department (ED) utilization will be assessed using the Emergency Department Information Exchange (EDIE) .
Time Frame: 6 months
Population: Data was unable to be obtained during the funding period. No data collection of EDIE utilization occurred during this study because team was unable to access EDIE data.
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Study reviewed by the University of Washington as minimal risk. Data Safety Monitoring Board (DSMB) not required by the funder or the University of Washington. Systematic assessment of SAE/AE or all-cause mortality not required by the funder or the University of Washington.
Arm/Group | ED-LINC Intervention Condition | Usual Care Condition
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03699085/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03699085/SAP_001.pdf